CLINICAL TRIAL: NCT03005756
Title: Single Center and Exploratory Investigator-initiated Trial to Evaluate the Safety and Efficacy of Needle Guiding Robot System for Radiofrequency Ablation in Hepatocellular Carcinoma Patients
Brief Title: Needle Guiding Robot for Radiofrequency Ablation: Safety and Efficacy Study on Hepatocellular Carcinoma Patients
Acronym: NGR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government); Hyundai Heavy Industries (Unknown)
Responsible Party: Principal Investigator, Hyung Jin Won, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Robin_RFA_01
Record Dates: First submitted 2016-12-26; First posted 2016-12-29 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot-assisted Radiofrequency Ablation (Experimental): CT-guided radiofrequency ablation of hepatocellular carcinoma using needle guiding robot
  Interventions: Device: Needle guiding robot

INTERVENTIONS:
Device: Needle guiding robot — This intervention is to evaluate the safety and efficacy of a needle guiding robot for assisting targeting in CT-guided radiofrequency ablation of hepatocelluar carcinomas.

SUMMARY:
The needle guiding robot helps targeting of radiofrequency ablation needles by matching computed tomography images and patients' bodies. Actual insertion of needles will be performed by doctors. This study evaluates the safety and efficacy of needle targeting on patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
A robotic system has been developed that includes a needle-path planning system and a needle-guiding robot arm with computed tomography (CT) guidance. The robot consists of robot base, 5-axis robot arm with guiding end-effector and path-planner. Optical tracking system with a custom-designed registration jig is used for the spatial registration and validation. Advantages of the robotic system would be accurate targeting with diverse angulation of the robot arm in CT-guided tumor ablation. Furthermore, robotic intervention might potentially decrease procedure time and radiation exposure to patients. The purpose of this clinical trial with patients with hepatocelluar carcinoma is to assess the safety and efficacy of our CT-guided needle-guiding robot.

ELIGIBILITY:
Inclusion Criteria:

* Patients with up to three Hepatocellular carcinomas (HCC) with no single HCC larger than 3 cm
* Candidates for CT-guided radiofrequency ablation of HCC
* Child-Pugh class A or B

Exclusion Criteria:

* Patients with untreatable/unmanageable coagulopathy
* Patients who are allergic to CT contrast media
* Patients with vascular invasion or extrahepatic metastases

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Total radiation exposure (DLP, mGy*cm) | At time of radiofrequency ablation
  Sum of radiation exposures measured during the radiofrequency ablation

SECONDARY OUTCOMES:
Number of repositioning of radiofrequency electrode | At time of radiofrequency ablation
  Number of repositioning of radiofrequency electrode in order to correct targeting discrepancy untile properly placed in to the target tumor
Targeting error | At time of the 1st insertion of the electrode
  Distance between the target and the electrode tip
Procedure time | At time of radiofrequency ablation
  Total period of time from the installation of needle guiding robot to patient's transfer after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koethe Y, Xu S, Velusamy G, Wood BJ, Venkatesan AM. Accuracy and efficacy of percutaneous biopsy and ablation using robotic assistance under computed tomography guidance: a phantom study. Eur Radiol. 2014 Mar;24(3):723-30. doi: 10.1007/s00330-013-3056-y. Epub 2013 Nov 13. PMID 24220755
- [Background] Abdullah BJ, Yeong CH, Goh KL, Yoong BK, Ho GF, Yim CC, Kulkarni A. Robot-assisted radiofrequency ablation of primary and secondary liver tumours: early experience. Eur Radiol. 2014 Jan;24(1):79-85. doi: 10.1007/s00330-013-2979-7. Epub 2013 Aug 9. PMID 23928933
- [Background] Abdullah BJ, Yeong CH, Goh KL, Yoong BK, Ho GF, Yim CC, Kulkarni A. Robotic-assisted thermal ablation of liver tumours. Eur Radiol. 2015 Jan;25(1):246-57. doi: 10.1007/s00330-014-3391-7. Epub 2014 Sep 5. PMID 25189152